CLINICAL TRIAL: NCT06465875
Title: The Effect of Book Reading on Comfort, Hope, Anxiety and Vital Signs of Intensive Care Unit Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Sevda Korkut, Associate Prof., TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024/147
Record Dates: First submitted 2024-06-09; First posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Hope; Comfort; Anxiety; Vital Signs
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will be read a storybook for three nights outside the routine practices of the clinic.
  Interventions: Other: Reading a book
- Control group (No Intervention): The control group will not be subjected to any practice other than the routine practices of the clinic.

INTERVENTIONS:
Other: Reading a book — Individuals in the intervention group will be read a storybook for three nights.
  Arms: Intervention group

SUMMARY:
This study was planned to investigate the effect of reading aloud books on comfort, hope, anxiety and vital signs in patients hospitalized in intensive care unit. This study was designed as a randomized controlled clinical trial. Data will be collected by using the Descriptive Characteristics Questionnaire, General Comfort Scale, Dispositional Hope Scale, State-Trait Anxiety Inventory, and the Vital Signs Monitoring Form.

DETAILED DESCRIPTION:
This study was planned to investigate the effect of reading aloud books on comfort, hope, anxiety and vital signs in patients hospitalized in intensive care unit. This study was designed as a randomized controlled clinical trial. Data will be collected by using the Descriptive Characteristics Questionnaire, General Comfort Scale, Dispositional Hope Scale, State-Trait Anxiety Inventory, and the Vital Signs Monitoring Form. Individuals in the intervention group will be read a storybook for 3 nights in the intensive care unit. The control group will not be subjected to any practice other than the routine practices of the clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years of age,
2. Stable clinical condition after intensive care unit admission,
3. Have no physical or mental impairment in answering the questions,
4. No verbal communication disability (hearing and speech),
5. No diagnosed psychiatric disorder,
6. With a Glasgow Coma Scale score of 15,
7. Not receiving sedation for at least 12 hours,
8. Will be hospitalized for at least 3 days from the time of enrollment in the study,
9. Individuals who agree to participate in the study will be included in the study.

Exclusion Criteria:

1. People with hearing or vision problems,
2. Intubated,
3. Any diagnosed neurological or psychological disorder,
4. Transferred to another unit or exitus before the specified period,
5. Individuals who do not agree to participate in the study will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Comfort level to be evaluated with the General Comfort Scale | After reading the book of the 3rd day
  It was developed to assess the comfort level of patients. The scale consists of three levels: relief, relaxation and superiority and four dimensions: physical, psychospiritual, sociocultural and environmental.
Level of hope to be assessed with the Dispositional Hope Scale | After reading the book of the 3rd day
  It was conducted to evaluate individuals' hope levels. It is an eight-point Likert type scale consisting of 12 items. Scores from the scale vary between 8 and 64.
Anxiety level to be assessed with State-Trait Anxiety Inventory | After reading the book of the 3rd day
  The inventory was developed to determine the state and trait anxiety levels of individuals. The scale consists of 40 items in total. While the first 20 items measure the state anxiety level, the items from 21 to 40 measure the trait anxiety level of the individual. The total score value obtained from both parts varies between 20 and 80.

SECONDARY OUTCOMES:
Blood pressure to be assessed with monitor | After reading the book of the 3rd day
  The patient's blood pressure will be measured from the brachial artery with a bedside monitor and the result will be recorded in mmHg.
Pulse to be assessed with monitor | After reading the book of the 3rd day
  Heart rate will be measured with a bedside monitor that can be measured from a finger and recorded as beats/min.
Oxygen saturation to be assessed with Pulse Oximeter | After reading the book of the 3rd day
  Oxygen saturation from the finger will be measured and recorded with a Pulse Oximeter.
Pain to be assessed with Numeric Rating Scale | After reading the book of the 3rd day
  The number "0" on the scale means that they do not feel any pain and the number "10" refers to the worst pain.

IPD SHARING:
Plan to Share IPD: No